CLINICAL TRIAL: NCT06489340
Title: A Phase 2a Open Label Study to Evaluate Cholesterol Efflux Mediator™ VAR200: 2- Hydroxypropyl-β-cyclodextrin (2-HPβCD) in Subjects With Type 2 Diabetic Kidney Disease (DKD)
Brief Title: P2a Open Label Study to Evaluate 2-HPβCD in Subjects With Diabetic Kidney Disease
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn due to patient enrollment challenges
Sponsor: ZyVersa Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VAR200-0301
Record Dates: First submitted 2024-06-18; First posted 2024-07-05 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-09

CONDITIONS: Diabetic Kidney Disease
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 2HPβCD (Experimental): Study drug will be administered by IV infusion during the treatment period.
  Interventions: Drug: 2HPβCD

INTERVENTIONS:
Drug: 2HPβCD — 2HPβCD is a 7 D-glucopyranosyl derivation of cyclodextrin (CD) that entraps and passively removes intracellular cholesterol from the kidney. It is also believed to promote active cholesterol removal through up-regulation of cholesterol efflux transporters ABCA1 and ABCG1.
  Other Names: 2-hydroxypropyl-β-cyclodextrin

SUMMARY:
This is an open label, two to three center study to evaluate the clinical efficacy and safety of 1 dose level of 2-hydroxypropyl-β-cyclodextrin (2-HPβCD) given intravenously in adult patients with type 2 diabetes with diabetic kidney disease (DKD) and proteinuria.

DETAILED DESCRIPTION:
This is a Phase 2a, open label, two to three center study to evaluate the clinical efficacy and safety of 1 dose level of 2-hydroxypropyl-β-cyclodextrin (2-HPβCD) given intravenously in adult patients with type 2 diabetes with diabetic kidney disease (DKD) and proteinuria.

The study will be conducted at 2 - 3 sites in the United States of America (USA) and will screen a sufficient number of subjects to complete 8 participants meeting the inclusion/exclusion criteria outlined.

The study consists of up to a 4-week screening period, a 12-week treatment period and a 4-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving and has provided a signed Informed Consent Form (ICF).
2. Male or female age 18 to 75 years inclusive, at the time of signing the informed consent.
3. Women of childbearing potential (WOCBP) and male subjects who are partners of WOCBP must agree to use an acceptable form of contraception during the study and for 30 days following the last dose of study drug.
4. Clinical diagnosis of type 2 diabetes as per guidelines.
5. Clinical diagnosis of diabetic kidney disease in the opinion of the principal investigator, or renal biopsy proven diabetic kidney disease without evidence of additional pathologic findings of alternative diagnosis.

   1. At screening, based on two 24-hour urine collections, geometric mean of two urinary albumin creatine ratios (UACR) ≥ 400 mg/g and ≤ 3500 mg/g.
   2. At screening, eGFR equal or greater than 30 and less than 90 mL/min/1.73 m^2.
6. Body mass index (BMI) ≤ 40.0 kg/m^2.
7. If on diabetes and anti-hypertensive medications:

   1. Angiotensin converting enzyme inhibitor (ACEi) or angiotensin receptor blocker (ARB) inhibitors dose must be stable for 3 months before screening.
   2. Sodium-glucose co-transporter 2 (SGLT2) or GLP-1 receptor agonist or long-acting insulin dose must be stable for at least 3 months prior to screening.
   3. All other diabetes and anti-hypertensive medications must be at a stable dose for at least 3 months prior to screening.
8. Hemoglobin A1c (HbA1c) ≤10.0% at screening.
9. Willing to comply with IV administration of the study drug for 12 weeks and all protocol procedures during the study.

Exclusion Criteria:

1. Has a solitary kidney.
2. Has a positive drug screen.
3. Known kidney disease other than diabetic kidney disease.
4. End stage renal disease (ESRD) (i.e., peritoneal dialysis, hemodialysis, or history of kidney transplantation).
5. Acute kidney injury or dialysis within the last 3 months before the screening visit.
6. Uncontrolled diabetes as defined by HbA1c >10 at screening.
7. Uncontrolled hypertension with systolic blood pressure (SBP) >140 mmHg or diastolic blood pressure (DBP) >90 mmHg during screening.
8. Unstable cardiovascular disease or history of myocardial infarction or arterial thromboembolic events within 3 months prior to screening or severe or unstable angina, New York Heart Association (NYHA) Class III or IV disease, or a QTc interval >480 msec.
9. Patients on IV medication containing cyclodextrin.
10. Patients on steroids, except for those on low-dose topical steroids (per PI discretion) or intranasal or inhaled steroids.
11. Surgery within the past 3 months prior to the first study drug administration determined by the Investigator to be clinically relevant.
12. Known malignancy that is progressing or has required active treatment within the past 3 years. Any exceptions must be approved by the Medical Monitor.

    a. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
13. Known history of Human Immunodeficiency Virus (HIV) infection (HIV 1/2 antibodies).
14. Known active Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection.
15. Diabetic ketosis, ketoacidosis and severe infections within a month or active infection requiring systemic therapy.
16. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participants' participation for the full duration of the study, or is not in the best interest of the participants to participate in the opinion of the treating Investigator.
17. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.
18. Women participants who are pregnant or breastfeeding or expecting to conceive children within the projected duration of the study or within 30 days of participation.
19. Aspartate aminotransferase (AST) or alanine transaminase (ALT) >3 upper limit of normal (ULN). One repeat test may be allowed within 7 days at the discretion of the Investigator.
20. Absolute neutrophil count ≤ 1.5 x 109/L at screening.
21. Platelets ≤ 100 x 109/L at screening.
22. Abnormal Hemoglobin (Hgb) (for men, abnormal levels are defined as <11.0 grams per deciliter (gm/dL) or >17.5 gm/dL. For women, < 10.0 gm/dL or >15.3 gm/dL.)
23. Currently participating or have participated in a study of an investigational product or used an investigational device within 3 months (or > 3 half-lives for mAbs with prolonged half-life of greater than 30 days) prior to the first dose of study intervention.
24. Patients on antibody therapeutics.
25. History or presence of alcohol or drug abuse within the 1 year prior to the first study drug administration.
26. A known history of otologic disease (e.g., Meniere's, sudden hearing loss, fluctuating hearing loss, vestibular schwannoma).
27. Pure tone air conduction thresholds in either ear at 3 consecutive frequencies > 60 dB at: 0.25, 0.5, 1, 2, 3, 4, 6, and 8 kHz.
28. Pure tone bone conduction thresholds > 60 dB in either ear that are 10 dB better than air conduction thresholds (i.e., air-bone gap > 10 dB) at all of the following frequencies: 0.5, 1, 2, and 4 kHz.
29. Use of non-steroidal anti-inflammatory drugs (NSAIDS) during the study period other than chronic low dose of aspirin stable for at least 3 months.
30. History of participation in a stem cell or gene therapy trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-06-11 (Actual); Primary Completion 2026-08-11 (Estimated); Study Completion 2026-08-11 (Estimated)

PRIMARY OUTCOMES:
Percent change in 24-hour urinary albumin to creatinine ratio (UACR) | From Day 1 (baseline) to Week 12 (end of treatment)
  Percentage change in urinary albumin to creatinine ratio (UACR) from baseline (day 1) to Week 12.
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | 12 Weeks
  Number of adverse events (AEs), serious adverse events (SAEs), discontinuations over the 12-week treatment period

SECONDARY OUTCOMES:
Absolute change in 24-hour urinary albumin to creatinine ratio (UACR) | From Day 1 (baseline) to Week 12 (end of treatment)
  Absolute change in 24-hour urinary protein to creatinine ratio (UPCR) from baseline (Day 1) to Week 12 (end of treatment)
Absolute change in 24-hour urinary protein to creatinine ratio (UPCR) | From Day 1 (baseline) to Week 12 (end of treatment)
  Absolute change in log transformed 24 hour urinary protein to creatinine ratio (UPCR) from Day 1 (baseline) to Week 12 (end of treatment)
Population trough pharmacokinetics of 2-hydroxypropyl-β-cyclodextrin (2-HPβCD) | Day 1, Day 29, Day 57, Day 85
  Trough plasma concentration of 2-hydroxypropyl-β-cyclodextrin (2-HPβCD) on Day 1, Day 29, Day 57, and Day 85, compared with pre-dosing concentrations on Day 1 and Day 4
Effects of 2-HPβCD on hearing based on changes in pure tone air conduction threshold from Day 1 to Week 16, and percent changes in tinnitus, and sense of fullness or stuffiness in the ears based on a Hearing Monitoring Questionnaire | From Day 1 to Week 16
  Changes in pure tone air conduction threshold based on audiometry testing from Day 1 to Week 16. Percent changes in the presence of tinnitus (ringing in the ears), and a sense of fullness or stuffiness in the ears based on responses to a Hearing Monitoring Questionnaire from Day 1 to Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Pergola, M.D PHD, Principal Investigator — Clinical Advancement Center, PLLC
Locations (1):
- Clinical Advancement Center, PLLC, San Antonio, Texas, United States